CLINICAL TRIAL: NCT04590144
Title: Safety and Performance of INVICTA Ventricular DF4 LEADS With Active Fixation-(APOLLO)
Acronym: APOLLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LINI01
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Ventricular Arrythmia; Lead; ICD; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: INVICTA lead
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- INVICTA lead (Experimental): All patients eligible for enrolment in whom the INVICTA lead is attempted (Implant of the INVICTA lead
  Interventions: Device: INVICTA lead

INTERVENTIONS:
Device: INVICTA lead — The implant or the attempt to implant an INVICTA lead
  Other Names: Implant of the INVICTA lead

SUMMARY:
The primary objective of this study is to assess the safety and key electrical performance of the INVICTA leads equipped with DF4 connector: ACTIVE fixation type models (single and dual coil: INVICTA 1CR, INVICTA 2CR)

DETAILED DESCRIPTION:
APOLLO study is a pre-market approval (INVICTA leads - devices under investigation - are not CE marked), interventional, prospective, longitudinal, international (European), multicenter, single arm study.

The devices under investigation, the INVICTA defibrillation leads, are new quadripolar leads, to be used with Implantable Cardiac Defibrillators and Cardiac Resynchronization Therapy Defibrillators (ICD/CRT-D).

This clinical study intends to demonstrate safety and electrical performances of the INVICTA leads among the different models: active fixation either single coil (model 1CR) or dual coil (model 2CR)leads models. The clinical data will be used to support the application to CE marking of INVICTA leads.

The primary endpoints will be evaluated at 3 months post-implantation; secondary endpoints will be evaluated up to 2 years post-implantation.

A total number of 445 patients will be enrolled in the study, in up to 60 centers in Europe.

The follow-up visits are scheduled at hospital discharge, at 1 month, at 3 months, at 6 months, at 12 months, at 18 months and at 24 months, post-implant

ELIGIBILITY:
Inclusion Criteria:

1. Any patient presenting an ICD or CRT-D indication as detailed in the latest ESC guidelines
2. Scheduled for a de-novo implant of an ICD (VR, DR) or CRT-D, manufactured by MicroPort CRM and equipped with a DF4 connector
3. Signed and dated informed consent

Exclusion Criteria:

1. Tricuspid valvular disease or any type of tricuspid replacement heart valve (mechanical or tissue)
2. Transient tachyarrhythmias due to reversible causes (such as drug intoxication, electrolyte imbalance, sepsis, hypoxia or other factors as myocardial infarction or electric shock)
3. Contraindication to a maximum single dose of 330 µg dexamethasone sodium phosphate (DSP)
4. Active myocarditis
5. Previous implant of pacemaker, ICD or CRT-D device and leads
6. Currently enrolled or planning to participate in a potentially confounding drug or device trial during the course of this study
7. Incapacitated subject or under guardianship, inability to understand the purpose of the study, or to meet follow-up visits at the implanting centre as defined in the investigational plan
8. Minor subjects
9. Pre-menopausal women
10. Drug addiction or abuse
11. Life expectancy less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
1.Freedom from INVICTA lead-related complications 1.Freedom from INVICTA lead-related complications [Time Frame: 90 days | 90 days
  Freedom from INVICTA lead-related complications as assessed by an independent events adjudicator and defined as any INVICTA lead-related serious adverse device effect (SADE) that resulted in patient death or required an additional invasive intervention
2.INVICTA lead electrical performance at 3 months | 3 months
  Right Ventricular (RV) pacing threshold (V) of the INVICTA lead, measured by the implanted ICD/CRT-D with 0.5 ms pulse width

SECONDARY OUTCOMES:
INVICTA lead pacing threshold | 24 months
  RV lead pacing threshold amplitude (V), measured by the implanted ICD/CRT-D with 0.5 ms pulse width
INVICTA lead impedances | 24 months
  RV lead pacing impedance (Ohm) and defibrillation coil impedance (Ohm), measured by the implanted ICD/CRT-D
INVICTA sensing threshold | 24 months
  RV lead endocardial R wave amplitude (mV), measured by the implanted ICD/CRT-D
Percentage of the shocks that successfully terminate a ventricular arrhythmia episode | 24 months
  Percentage of endocardial shock therapies that successfully terminate ventricular arrhythmia episodes, calculated as the proportion of successful shocks on the total number of shocks delivered during defibrillation testing or spontaneous ventricular arrhythmias
Acute INVICTA lead complications | 30 days
  Assessment of Acute INVICTA lead complications
Chronic INVICTA lead complications | > 30 days
  Assessment of Chronic INVICTA lead complications
Daily INVICTA autothreshold values (V) | 1 month
  Assessment of Daily INVICTA autothreshold values (V)
.INVICTA lead handling assessment | At implant (day 0)
  Summary of the investigators' opinion about INVICTA handling at implant
INVICTA lead implant success rate | At implant (day 0)
  % of enrolled patients successfully implanted with an INVICTA lead
Serious Adverse Events up to 24 months | 24 months
  Report of SAEs occurred up to 24 months post-implantation

OTHER OUTCOMES:
Acute complication rates as a function of the lead position | < 30 days
  Acute complication rates as a function of the lead position (apical vs septal)
Chronic complication rates as a function of the lead position | > 30 days
  Chronic complication rates as a function of the lead position (apical vs septal
Electrical performances as a function of the lead position | 24 months
  Electrical performances as a function of the lead position (apical vs septal)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Marques, MD, Principal Investigator — Hospital de Santa Maria - Lisboa - Portugal
Locations (45):
- Kepler Universitätsklinikum GmbH, Linz, Austria
- France (8):
  - CH Annecy, Annecy
  - CHU Brest, Brest
  - CHU Clermont- Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - CHU Lille, Lille
  - Hôpital St Joseph, Marseille
  - CHU Strasbourg, Strasbourg
  - CHU Tours, Tours
- Germany (5):
  - RWTH Aachen, Aachen
  - Herz- und Gefäßzentrum Bad Bevensen, Bad Bevensen
  - Evangelisches Klinikum Bethel, Bielefeld
  - Universitäts- Herzzentrum Freiburg -Bad Krozingen, Freiburg im Breisgau
  - Hausärztlich- Kardiologisches MVZ "Am Felsenkeller" GmbH, Pirna
- Italy (8):
  - Cliniche Humanitas Gavazzeni, Bergamo
  - Ospedale di Desenzano del Garda, Desenzano del Garda
  - Ospedale Piemonte (IRCCS Bonino Pulejo), Messina
  - AO di Rilievo Nazionale A. Cardarelli, Napoli
  - Univ. degli Studi della Campania L. Vanvitelli, Napoli
  - Osp SS Annunziata, Taranto
  - AO Univ. S. Maria della Misericordia, Udine
  - AULSS 8 Berica - Vicenza, Vicenza
- Netherlands (2):
  - Elisabeth Tweesteden Ziekenhuis, Tilburg
  - Isala Klinieken, Zwolle
- Portugal (8):
  - ULS Amadora/Sintra, Amadora
  - ULS de Coimbra, Coimbra
  - ULS do Alto Ave, Creixomil
  - ULS Alentejo Central, Evora
  - Hospital Santa Maria, Lisbon
  - ULS de Sao Jose - Hospital Santa Marta, Lisbon
  - ULS Santo Antonio, Porto
  - ULS Gaia/Espinho, Vila Nova de Gaia
- Spain (10):
  - Hospital Clínico Universitario de Valencia, Valencia, Spain
  - Hospital General de Alicante, Alicante
  - Hospital Josep Trueta,, Girona
  - Hospital Virgen de las Nieves, Granda
  - Hospital Universitario de Gran Canaria, Las Palmas
  - Hospital Clinico de Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
- United Kingdom (3):
  - Barnet Hospital, Royal Free Trust, Barnet
  - Queen Elizabeth, Birmingham
  - Great Western Hospital, Swindon